CLINICAL TRIAL: NCT03634462
Title: Complete Decongestive Therapy With Negative Pressure for Lipedema and Lymphedema Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Lipedema Foundation (Other)
Responsible Party: Principal Investigator, Manus Donahue, Associate Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160199; LF Award #12 (Other Grant/Funding Number: Lipedema Foundation)
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Lipedema; Secondary Lymphedema
Keywords: lipedema; lymphedema; therapy; sodium; swelling
MeSH Terms: conditions — Lipedema; Lymphedema | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Intervention Model Description: Subjects with lipedema or secondary leg lymphedema will receive standard manual lymphatic drainage therapy with negative pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Lipedema (Experimental): Females with lipedema who meet the inclusion and exclusion criteria for lipedema and this study requirements. The intervention in this arm is a course of CDT with graded negative pressure.
  Interventions: Other: CDT with graded negative pressure
- Patients with secondary leg lymphedema (Experimental): Patients with secondary leg lymphedema following cancer therapies will be limited to the female gender since the comparison group of patients have lipedema which is a condition predominantly effecting females. These patient subjects will consist of those who meet the inclusion and exclusion criteria for secondary leg lymphedema and this study requirements. The intervention in this arm is a course of CDT with graded negative pressure.
  Interventions: Other: CDT with graded negative pressure

INTERVENTIONS:
Other: CDT with graded negative pressure — Complete Decongestive Therapy (CDT)is a common conservative intervention involving stimulation of the lymphatic system, use of compression, skin care and exercise. The use of graded negative pressure in conjunction with CDT is another conservative therapy intervention used to help clear the lymphatic congestion.

SUMMARY:
This study is designed to investigate the therapy outcomes from routine physical therapy in persons with lipedema and secondary limb lymphedema. Complete decongestive therapy (CDT) is a common conservative treatment to optimize lymphatic functioning using exercise, compression, lymphatic stimulation and skin care. PhysioTouch is a gentle graded negative pressure device designed to enhance lymphatic stimulation that is used by the skilled therapist in conjunction with hands on techniques of tissue mobilization for enhanced clearance of lymph stasis in persons with lymphedema. This study will investigate the conservative treatment impact in patients with lipedema and lower extremity lymphedema using this conservative available technique.

DETAILED DESCRIPTION:
This study will assess the treatment impact of complete decongestive therapy (CDT) in conjunction with negative pressure application using PhysioTouch (R) in women with lipedema or secondary lymphedema. Lipedema is an adipose tissue disorder in which persons experience pain and swelling in their legs and lower quadrants. Lipedema is a disorder that almost exclusively effects females, is frequently inherited, and is triggered by hormonal changes. Symptomatology includes symmetric swelling of the hypodermis of the legs, indentations in the fat causing uneven skin which may include large extruding mounds of tissue, is often accompanied by lymphedema, and is unresponsive to diet or exercise.

Women with secondary limb lymphedema in this study are persons who have developed lymphedema following cancer treatment. Persons with lymphedema or lipedema often receive CDT. CDT is a common conservative treatment to optimize lymphatic functioning using exercise, compression, lymphatic stimulation and skin care. An adjunct component of therapy is the use of gentle graded negative pressure to further enhance lymphatic stimulation. PhysioTouch is a gentle graded negative pressure device designed to enhance lymphatic stimulation.

The investigators will evaluate to what extent CDT with graded negative pressure impacts lymphatic functioning in patients with lipedema or lymphedema of the lower extremities. Additionally, the investigators will also noninvasively evaluate lymphatic function using Magnetic Resonance (MR) lymphangiography without contrast, and whether tissue sodium and fat composition are associated with reduced lymphatic pumping dynamics in the study's group cohorts. This will provide new information on the mechanism of dysfunctional fat clearance in patients with lipedema using traditional conservative therapy. By outlining internal mechanisms underlying lipedema etiology, and their response to CDT, this will provide objective markers elucidating the unique characteristics of lipedema compared with secondary lymphedema.

Study hypothesis: Therapeutic manipulation of lymphatic stasis over six weeks increases lymphatic pumping kinetics and reduces tissue sodium accumulation.

Biophysical measurements will also be acquired, including bioimpedance spectroscopy and perometry. Three cohorts will be studied: age-, gender-, and BMI-matched study controls, patients with lipedema, and patients with secondary unilateral leg lymphedema from cancer therapies. Only females will be recruited since lipedema primarily affects females. Only patients with leg lymphedema following cancer therapies will be recruited to control for the known reason for leg lymphedema. Subjects will be recruited from age 14 years and older since lipedema is triggered by hormonal changes occurring with menarche and pregnancy. Measurements will be repeated on a separate study date in a subset of volunteers. Reproducibility will be determined using an intraclass correlation coefficient; results will establish the normative range of these measures in healthy tissue. Significant differences in imaging metrics and biophysical measures between groups will be evaluated using a one-way ANOVA. This work will improve the investigators understanding of the physiology of lipedema compared to obesity and lymphedema. The results will determine the potential for these measures to serve as biomarkers of lipedema, as distinguished from obesity or on a spectrum of lymphedema. The results will also evaluate for changes in lymphatic pumping and tissue sodium accumulation following a commonly used physical therapy intervention over a course of 6 weeks in the two patient populations, lipedema (n=5) and secondary leg lymphedema (n=5).

ELIGIBILITY:
Inclusion Criteria:

* Females with a diagnosis of lipedema or a probable diagnosis of lipedema
* Females with a diagnosis of secondary limb lymphedema following cancer treatments

Exclusion Criteria:

* Subjects who have any type of non-MRI compatible bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.) or are not able to comfortably be able to tolerate the limited fit of the MRI
* Subjects who have any type of ferromagnetic bioimplant that could potentially be displaced.
* Subjects who may have shrapnel imbedded in their bodies (such as from war wounds), metal workers and machinists (potential for metallic fragments in or near the eyes).
* Pregnant women will be excluded from the MRI portion of the study only
* Subjects who have open wounds on either ankle or top of foot because of contraindications with placement of electrodes to obtain the L-DEX U400 readings.
* Persons with heart pacemakers.
* Persons with Dercum's disease, diabetes or high blood pressure (systolic great than 140 and diastolic great than 90).

Ages: 14 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Assessing a Change in Bioimpedance Spectroscopy (BIS) Following CDT with Graded Negative Pressure | At baseline and at 6-8 weeks following the completion of therapy
  BIS quantified using Impedimed L-dex

SECONDARY OUTCOMES:
Assessing a Change in Lymphatic stasis Following CDT with Graded Negative Pressure | At baseline and at 6-8 weeks following the completion of therapy
  Quantitative analysis of lymphatic stasis using non-invasive MR lymphangiography
Assessing a Change in Limb Volume Following CDT with Graded Negative Pressure | At baseline and at 6-8 weeks following the completion of therapy
  Volume quantified using Perometer
Assessing a Change in Sodium Levels in Regions of Interest Following CDT with Graded Negative Pressure | At baseline and at 6-8 weeks following the completion of therapy
  Quantitative analysis of sodium levels using non-invasive sodium MRI

CONTACTS AND LOCATIONS:
Overall Officials: Manus J Donahue, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crescenzi R, Marton A, Donahue PMC, Mahany HB, Lants SK, Wang P, Beckman JA, Donahue MJ, Titze J. Tissue Sodium Content is Elevated in the Skin and Subcutaneous Adipose Tissue in Women with Lipedema. Obesity (Silver Spring). 2018 Feb;26(2):310-317. doi: 10.1002/oby.22090. Epub 2017 Dec 27. PMID 29280322